CLINICAL TRIAL: NCT01189136
Title: Percutaneous Posterior Tibial Nerve Stimulation for the Treatment of Acute Postoperative Voiding Dysfunction
Brief Title: Treatment for Acute Postoperative Voiding Dysfunction
Acronym: PTNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Charles Rardin, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-0061; 06-0061 (Other: WIHRI)
Record Dates: First submitted 2010-08-20; First posted 2010-08-26 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Urinary Retention
Keywords: Voiding dysfunction
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham treatment (Sham Comparator): 34 gauge needle inserted 3cm above the medial ankle, but nonconductive cables are connected, so that no electrical stimulation is applied, over a 30-minute treatment period
  Interventions: Other: Sham treatment
- PTNS Active Treatment (Experimental): 34 gauge needle inserted 3cm above the medial ankle, and cables are connected to the PTNS stimulator device. Stimulation is provided, per manufacturer directions, over a 30-minute treatment period
  Interventions: Device: PTNS Active Treatment

INTERVENTIONS:
Device: PTNS Active Treatment — 34 gauge needle inserted 3cm above the medial ankle, and cables are connected to the PTNS stimulator device. Stimulation is provided, per manufacturer directions, over a 30-minute treatment period.
  Arms: PTNS Active Treatment
Other: Sham treatment — 34 gauge needle inserted 3cm above the medial ankle, but nonconductive cables are connected, so that no electrical stimulation is applied, over a 30-minute treatment period
  Arms: Sham treatment

SUMMARY:
If patients are unable to have their foley catheter removed because their bladder is not emptying well, they may be eligible for study participation. This study is designed to evaluate whether Posterior Tibial Nerve Stimulation is effective in improving bladdder function after surgery. Study participation is limited to one day.

DETAILED DESCRIPTION:
If patients fail a voiding trial (the test done to see if a foley catheter is ready to be removed after surgery), they may be offered participation in this trial. Patients are randomized to receive active treatment or a sham treatment. A small, accupuncture-type needle is inserted through the skin just above the ankle. A small, battery-powered generator will be attached to the needle. The generator will give a low-voltabe stimulation which is adjusted for comfort level and applied for 30 minutes. After treatemnt, the voiding trial will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* First voiding trial after Urogynecological surgery shows that bladder is not emptying well.

Exclusion Criteria:

* Patient declines participation.

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Rardin, MD, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
No plans to make IPD available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 112 subjects invited to participate, 28 declined, and 84 were equally distributed between treatment and sham groups
Groups:
- Sham Treatment: No electrical stimulation is actually received
  Sham treatment: No electrical stimulation is given
- Peructaneous Tibial Nerve Stimulation: Patient receives PTNS for 30 minutes
  PTNS treatment: Electrical stimulation is received
Period: Overall Study
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 36 | 75
  >=65 years | 3 | 6 | 9
Age, Customized [Mean (Standard Deviation); unit: years] | 46 (8) | 54 (11) | 50 (9)
Gender [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 0 | 0 | 0
Parity [Mean (Standard Deviation); unit: pregnancies] | 2 (1) | 2 (1) | 2 (1)
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.0 (3.1) | 28.7 (3.5) | 28.9 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Persistent Retention
Description: Number of participants with persistent unsuccessful trial of void after the intervention
Time Frame: 30 minutes
Measure: Number; unit: participants
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Number analyzed (Participants) | 42 | 42
participants | 29 | 21

2. Secondary Outcome: Amount of Improvement in Voiding Efficiency
Description: Improvement of voiding efficiency, as measured by dividing the volume voided by the total volume (voided volume + retained volume) per participant. Each participant is evaluated separately, and the mean percentage of improvement was calculated for each arm.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of voided vol/total volume
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Number analyzed (Participants) | 42 | 42
percentage of voided vol/total volume | 21 (8) | 28 (5)

3. Other Pre Specified Outcome: Questionnaire Data - Impression of Allocation
Description: Participants were asked to guess to which treatment arm they had been allocated ("PTNS" "Sham" or "I Don't Know"). Outcome was measured as the number of patients in each arm accurately determining their allocation.
Time Frame: 30 minutes
Population: Number
Measure: Number; unit: number of participants
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Number analyzed (Participants) | 42 | 42
number of participants | 10 | 41

4. Other Pre Specified Outcome: Pain From Treatment
Description: Patient-reported discomfort attributable to the study intervention (0-10 Likert scale, with higher numbers representing greater pain)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Number analyzed (Participants) | 42 | 42
units on a scale | 0.14 (0.08) | 0.55 (0.09)

ADVERSE EVENTS:
Time Frame: 1 hour (30 minutes of treatment, then 30 minutes of observation prior to hospital discharge)
Description: Any adverse events were collected by the investigators.
Arm/Group | Sham Treatment | Peructaneous Tibial Nerve Stimulation
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No